CLINICAL TRIAL: NCT01572922
Title: Massive Iron Deposit Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Regional One Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIDAS; R01DK088988 (NIH)
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-04

CONDITIONS: Iron Overload; Excessive Body Iron Burden
Keywords: Sickle cell disease; Thalassemia; Hemochromatosis; Cancer
MeSH Terms: conditions — Iron Overload; Anemia, Sickle Cell; Thalassemia; Hemochromatosis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Iron-overloaded (Other): Patients with iron overload or excessive body iron burden, a serious condition resulting from increased dietary gastro¬intestinal absorption, multiple erythrocyte transfusions, or both.
  Interventions: R2*-UTE, R2*-GRE, and if clinically indicated, liver biopsy.
  Interventions: Device: R2*-UTE; Device: R2*-GRE; Procedure: Liver biopsy

INTERVENTIONS:
Device: R2*-UTE — Ultra short echo time (UTE) magnetic resonance imaging (MRI). Study participants will undergo an MRI examination of the liver on a 1.5T MRI and a 3T MRI scanner each. Because liver biopsy metal needle fragments could interfere with the MRI measurements, the MRI exams will always precede liver biopsy. Multi-echo GRE sequences will be used to acquire images with increasing TEs. Images of the liver will be obtained in transversal slice orientation through the center of the liver at the level of the origin of the main portal vein. At equivalent slice locations R2*-UTE scans will be performed.
Device: R2*-GRE — Gradient-echo (GRE) magnetic resonance imaging (MRI). Study participants will undergo an MRI examination of the liver on a 1.5T MRI and a 3T MRI scanner each. Because liver biopsy metal needle fragments could interfere with the MRI measurements, the MRI exams will always precede liver biopsy. Multi-echo GRE sequences will be used to acquire images with increasing TEs. Images of the liver will be obtained in transversal slice orientation through the center of the liver at the level of the origin of the main portal vein. At equivalent slice locations R2*-UTE scans will be performed.
Procedure: Liver biopsy — Indications for liver biopsy include, but are not limited, to the need to quantify liver tissue iron and the need to obtain histopathological information of the liver tissue. Liver biopsies will only be performed if clinically indicated and will be done only once per patient. The technique to be used is coaxial percutaneous (transcapsular) technique; however, a coaxial transjugular technique may be performed in subjects with increased bleeding diathesis, since it is associated with less hemorrhagic risk. Healthy volunteers will not undergo liver biopsy.

SUMMARY:
Iron overload is a severe complication of multiple blood transfusions. As the body has no physiologic mechanism for clearing iron, repeated transfusions cause iron accumulation in organs and lead to iron toxicity. Accurate assessment of iron overload is paramount to quantify excessive iron accumulation and to monitor response to iron chelation therapy. Magnetic resonance imaging (MRI) methods have been used to noninvasively measure hepatic iron concentration (HIC). Although MRI-based measurements of transverse relaxation rates (R2 and R2*) accurately predict biopsy-proven HICs below 15 mg Fe/g, previous studies have shown that their precision is limited for HICs above 15 mg Fe/g and inaccurate above 25 mg Fe/g. Current R2* gradient-echo (GRE) MR techniques fail occasionally for very high iron overloads (HIC ~ 15-25 mg Fe/g) and always for massive iron overloads (HIC > 25 mg Fe/g) because R2* is so high that the MR signal decays before it can be measured accurately.

Overall accrual: 200 patients

Purpose: To determine if a new MRI (UTE) can measure the amount of iron in the liver of people with large amounts of iron and compare the results with the same patient's liver bx. Estimated patient accrual is 150. It is estimated that 41 of these patients will have clinical indication for liver biopsy.

DETAILED DESCRIPTION:
The MIDAS study is a prospective and non-therapeutic study that will test a new MRI technique for the assessment of iron overload in the liver: the newly developed ultra short echo time (UTE), R2*-UTE. The R2*-UTE technique, developed by St. Jude investigators from the Department of Radiological Sciences, will be first tested in healthy volunteers for feasibility and implementation of the technique. The technique will then be tested in research participants, who will have both the R2*-GRE and the R2*-UTE techniques performed, in addition to a liver biopsy for liver iron quantitation if clinically indicated. Quantitation of liver tissue iron will be done at Mayo Clinic Laboratory in Rochester, Minnesota.

Primary Objective:

* To test the association of hepatic iron content (HIC) measured with the newly developed 1.5T R2*-UTE technique and HIC quantified by liver biopsy in subjects with iron overload.

Secondary Objectives:

* To explore the relationship between 1.5T R2*-UTE and 1.5T R2*-GRE measurements in subjects with iron overload.
* To explore the relationship between 1.5T R2*-UTE measurements with iron studies (serum iron and transferrin saturation) in subjects with iron.

ELIGIBILITY:
Inclusion Criteria

* History of 12 or more lifetime erythrocyte transfusions, AND
* Need for liver iron content assessment (by MRI or liver biopsy)

Exclusion Criteria

* Presence of certain MR-unsafe foreign material in the body, or other conditions that make the research participant ineligible for an MRI scan per St. Jude policies.
* Any condition or chronic illness that in the opinion of the PIs makes participation on study ill-advised.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hankins, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients within the St. Jude Network (St. Jude Children's Research Hospital, St. Jude Domestic Affiliates, and the adult Hematology and Oncology program at the University of Tennessee Health Sciences Center) who have history of 12 or more lifetime erythrocyte transfusions, and need for liver iron content assessment.
Pre-assignment Details: One arm study
Groups:
- Arm 1: All eligible patients with history of 12 or more lifetime erythrocyte transfusions, and need for liver iron content assessment.
Period: Overall Study
Arm/Group | Arm 1
Started | 142
Completed | 139
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 85
  Between 18 and 65 years | 57
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 15.9 [1.5 to 53.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 131
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10
  Black or African American | 85
  White | 40
  More than one race | 1
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Iron Content in the Liver Using Liver Biopsy
Description: Hepatic iron content in the liver using liver biopsy
Time Frame: up to 30 days after MRI
Population: Eligible iron-overloaded patients with both liver biopsy measurement and 1.5T R2*-UTE measurement.
Measure: Median (Full Range); unit: mcg
Groups:
- Iron-overloaded Patients: Eligible iron-overloaded patients with both liver biopsy measurement and 1.5T R2*-UTE measurement
Arm/Group | Iron-overloaded Patients
Number analyzed (Participants) | 41
mcg | 19.8 [0.1 to 45.0]

2. Primary Outcome: MRI-derived R2* Values Using 1.5T UTE Technique
Description: Hepatic iron content of the liver using MRI-derived 1.5T R2*-UTE measurement, with results in Hz. R2* is a measure obtained with MRI, i.e., MRI R2*. It is measured in hertz (Hz). In lay terms, the MRI machine picks up a signal back from the tissue during the process of scanning the tissues. With every "picture taken", this signal is strong in the beginning and then wanes off. R2* reflects how fast the signal wanes off. If there is too much iron in the tissue, the signal disappears faster, making the T2* value low. T2* is the reciprocal of R2* (R2*= 1/T2*). So, if the signal drops fast, the T2* is low and the R2* is high. In this study, we are measuring the R2* value. The higher the R2*, the more iron in the liver tissue. We can compare the R2* value with that of a liver biopsy to then use the R2* value to tell us how much iron is in the liver without having to biopsy the liver.
Time Frame: Up to 30 days after MRI
Population: Eligible iron-overloaded patients with both liver biopsy measurement and 1.5T R2*-UTE measurement.
Measure: Median (Full Range); unit: Hz
Arm/Group | Iron-overloaded Patients
Number analyzed (Participants) | 41
Hz | 864.4 [45.4 to 2245.5]

3. Secondary Outcome: MRI-derived R2* Using 1.5T GRE Technique
Description: MRI-derived R2* Using 1.5T GRE Technique in Hz. R2* is a measure obtained with MRI, i.e., MRI R2*. It is measured in hertz (Hz). In lay terms, the MRI machine picks up a signal back from the tissue during the process of scanning the tissues. With every "picture taken", this signal is strong in the beginning and then wanes off. R2* reflects how fast the signal wanes off. If there is too much iron in the tissue, the signal disappears faster, making the T2* value low. T2* is the reciprocal of R2* (R2*= 1/T2*). So, if the signal drops fast, the T2* is low and the R2* is high. In this study, we are measuring the R2* value. The higher the R2*, the more iron in the liver tissue. We can compare the R2* value with that of a liver biopsy to then use the R2* value to tell us how much iron is in the liver without having to biopsy the liver.
Time Frame: Up to 30 days after MRI
Population: Iron-overloaded patients had 1.5T R2*-GRE measurements.
Measure: Median (Full Range); unit: Hz
Groups:
- Iron-overloaded Patients: Iron-overloaded patients defined as having more than 12 transfusions in their lifetime as measured with R2* using 1.5T GRE.
Arm/Group | Iron-overloaded Patients
Number analyzed (Participants) | 139
Hz | 333.8 [33.6 to 2726.3]

4. Secondary Outcome: MRI Derived R2* Using 1.5T UTE Technique
Description: MRI-derived R2* value using 1.5T R2*-UTE in Hz. R2* is a measure obtained with MRI, i.e., MRI R2*. It is measured in hertz (Hz). In lay terms, the MRI machine picks up a signal back from the tissue during the process of scanning the tissues. With every "picture taken", this signal is strong in the beginning and then wanes off. R2* reflects how fast the signal wanes off. If there is too much iron in the tissue, the signal disappears faster, making the T2* value low. T2* is the reciprocal of R2* (R2*= 1/T2*). So, if the signal drops fast, the T2* is low and the R2* is high. In this study, we are measuring the R2* value. The higher the R2*, the more iron in the liver tissue. We can compare the R2* value with that of a liver biopsy to then use the R2* value to tell us how much iron is in the liver without having to biopsy the liver.
Time Frame: up to 30 days after MRI
Population: Iron-overloaded patients had 1.5T R2*-UTE-measurement.
Measure: Median (Full Range); unit: HZ
Groups:
- Iron-overloaded Patients: Iron-overloaded patients with R2* using 1.5T UTE
Arm/Group | Iron-overloaded Patients
Number analyzed (Participants) | 139
HZ | 319.2 [45.2 to 2245.5]

5. Secondary Outcome: R2* Using 1.5T UTE Technique for Patients With Serum Iron and Transferrin Saturation Measurements
Description: MRI-derived R2* value using 1.5T R2*-UTE in Hz for patients who have had serum iron and transferrin saturation measurements. R2* is a measure obtained with MRI, i.e., MRI R2*. It is measured in hertz (Hz). In lay terms, the MRI machine picks up a signal back from the tissue during the process of scanning the tissues. With every "picture taken", this signal is strong in the beginning and then wanes off. R2* reflects how fast the signal wanes off. If there is too much iron in the tissue, the signal disappears faster, making the T2* value low. T2* is the reciprocal of R2* (R2*= 1/T2*). So, if the signal drops fast, the T2* is low and the R2* is high. In this study, we are measuring the R2* value. The higher the R2*, the more iron in the liver tissue. We can compare the R2* value with that of a liver biopsy to then use the R2* value to tell us how much iron is in the liver without having to biopsy the liver.
Time Frame: Up to 30 days after MRI
Population: 1.5T R2*-UTE from eligible patients who had 1.5T R2*-UTE, serum iron, and transferrin saturation measurements.
Measure: Median (Full Range); unit: Hz
Arm/Group | Iron-overloaded Patients
Number analyzed (Participants) | 104
Hz | 340.8 [45.2 to 2245.5]

6. Secondary Outcome: Serum Iron Measurements Compared With 1.5T R2* UTE
Description: Serum iron measurements from eligible patients had 1.5T R2*-UTE and serum iron and transferrin saturation measurements.
Time Frame: Up to 30 days after MRI
Population: Iron-overloaded patients had 1.5T R2*-UTE and serum iron and transferrin saturation measurements.
Measure: Median (Full Range); unit: ug/dL
Groups:
- Serum Iron Measurements: Serum iron measurements from eligible patients had 1.5T R2*-UTE and serum iron and transferrin saturation measurements.
Arm/Group | Serum Iron Measurements
Number analyzed (Participants) | 104
ug/dL | 156.5 [35 to 311]

7. Secondary Outcome: Transferrin Saturation Measurements
Description: Iron Transferrin Saturation in % measurements Transferrin Saturation measurements from eligible patients had 1.5T R2*-UTE and serum iron and transferrin saturation measurements.
Time Frame: Up to 30 days after MRI
Population: Iron-overloaded patients had 1.5T R2*-UTE and serum iron and transferrin saturation measurements.
Measure: Median (Full Range); unit: percentage
Groups:
- Iron-overloaded Patients: Iron-overloaded patients with 1.5T R2*-UTE and serum iron and transferrin saturation measurements.
Arm/Group | Iron-overloaded Patients
Number analyzed (Participants) | 104
percentage | 71 [12 to 157]

ADVERSE EVENTS:
Time Frame: Time frame for adverse event reporting is 10 days following the last study procedure for eligible patients.
Arm/Group | Iron-overloaded Patients
All-Cause Mortality (participants affected / at risk) | 1/142
Serious Adverse Events (participants affected / at risk) | 1/142
Other Adverse Events (participants affected / at risk) | 2/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron-overloaded Patients (N=142)
Infections and infestations (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron-overloaded Patients (N=142)
Anxiety (Psychiatric disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT01572922/Prot_SAP_000.pdf